CLINICAL TRIAL: NCT06805552
Title: Prognostic Model of Survival of Patients With Hepatocarcinoma and Sarcopenia Treated With Systemic Therapy
Brief Title: Sarcopenia and Systemic Therapy in HCC
Acronym: Sarco HCC
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: Sarco HCC
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sarcopenia; HCC systemic therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC Patients: Patients with hepatocellular carcinoma treated with systemic therapy

SUMMARY:
This is a multi-center, retrospective observational study in patients with liver cancer (HCC) to assess the impact of sarcopenia (muscle loss) on the prognosis, duration, and tolerance of systemic treatment.

DETAILED DESCRIPTION:
The impact of sarcopenia will be assessed 12 months after the start of chemotherapy. Additionally, other factors affecting prognosis will be investigated to develop a specific predictive model for the risk of death at 12 months. Finally, an external validation of this predictive model for the risk of death will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Diagnosis of hepatocellular carcinoma based on histological and/or radiological results as defined by the European Association for the Study of the Liver (EASL) and the American Association for the Study of Liver Diseases (AASLD). The staging of hepatocellular carcinoma was obtained through contrast-enhanced liver CT and/or MRI.
* Patients with advanced (BCLC-C) or intermediate (BCLC-B) stage hepatocellular carcinoma, or patients with early-stage (BCLC-A) hepatocellular carcinoma who have not responded to previous locoregional ablative treatments and/or liver resection.
* Treatment with TKIs according to the indications and prescription criteria defined by AIFA, with no requirement to reach a minimum treatment period.

Availability of a CT scan performed within no more than 8 weeks prior to the start of TKI therapy.

- Obtaining written informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected with Hepatocellular Carcinoma
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of Sarcopenia in HCC patient's survival | From January 2008 to April 2021
  Evaluation of the prognostic role of sarcopenia in the survival of patients affected by HCC in liver cirrhosis and candidates for systemic treatment. Possible development of a specific classification system for the risk of death.

SECONDARY OUTCOMES:
Role of Sarcopenia in HCC systemic therapy tolerability | From January 2008 to April 2021
  Evaluation of the role of sarcopenia on the duration and tolerability of systemic treatment in patients affected by HCC in liver cirrhosis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS AOUBO Policlinico di S.Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No